CLINICAL TRIAL: NCT01422018
Title: Effect of Intravitreal Bevacizumab on Focal Edema With Hard Exudates Secondary to Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Won Ki Lee, Pf., Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC11MISI0439
Record Dates: First submitted 2011-08-05; First posted 2011-08-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Complications
Keywords: clinically significant macular edema; diabetic macular edema; focal edema; focal laser photocoagulation; hard exudates; intravitreal bevacizumab
MeSH Terms: conditions — Diabetes Complications | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm for Anastin injection (Experimental): intravitreal Avastin injection
  Interventions: Drug: Avastin (bevacizumab)

INTERVENTIONS:
Drug: Avastin (bevacizumab) — Bevacizumab (1.25 mg in 0.05 ml) (Avastin; Genentech Inc., San Francisco, CA, USA)

SUMMARY:
Purpose: To evaluate the efficacy of intravitreal bevacizumab (IVB) on focal edema with hard exudates secondary to diabetic retinopathy.

Design: Prospective interventional case series. Participants: Ten eyes of 10 consecutive patients showing focal edema with hard exudates secondary to diabetic retinopathy which are not eligible for focal laser photocoagulation due to central location (< 500 µm from fovea).

ELIGIBILITY:
Inclusion Criteria:

1. patients of either gender aged > 18 years
2. patients with type 2 diabetes
3. central macular thickness > 300 µm on OCT
4. eyes not eligible for focal laser photocoagulation due to the central location of hard exudates (< 500 µm)
5. an area of retinal thickening less than 2 disc areas in diameter
6. 67% or more of leakage associated with microaneurysms

Exclusion Criteria:

1. eyes with history of laser photocoagulation or pharmacological intervention for DME on study eye
2. eyes with any pharmacologic intervention on fellow eye within 6 months
3. history of ocular diseases other than diabetic retinopathy
4. surgical history other than cataract extraction with intraocular lens implantation
5. panretinal photocoagulation within 3 months of enrollment
6. media opacity
7. any thromboembolic event within 6 months, or evidence of active cardiac ischemia on electrocardiogram (ECG) at time of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Changes in best-corrected visual acuity (BCVA) | from month 0 to month 6 in monthly schedule (upto 6 months)
  ETDRS BCVA will be measured after 6 6 serial IVB.

SECONDARY OUTCOMES:
amount of hard exudates detected on fundus photography | from month 0 to month 6 in bimonthly schedule (upto 6 months)
  on fundus photography
macular edema detected by optical coherent tomography | from month 0 to month 6 in bimonthly schedule (upto 6 months)
  central subfield thickness will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Won ki Lee, MD Ph.D, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's hospital, Seocho, Seoul, South Korea